CLINICAL TRIAL: NCT02155036
Title: The Effect of Exercise on Renal Function and Cardiovascular Disease in Pre-dialysis (Chronic Kidney Disease Stage 3-4) Patients With Chronic Kidney Disease; a Randomised Controlled Trial Pilot Study.
Brief Title: Effect of Exercise on Renal Function in Predialysis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCH11-123
Record Dates: First submitted 2014-05-27; First posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Kidney Disease
Keywords: exercise; rehabilitation; kidney function; cardiovascular disease risk
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Usual care
- Exercise (Active Comparator): exercise intervention
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The intervention will include 2 sessions of gym-based exercise per week, both of which will be supervised for 3 months, supervision will then decrease to once-weekly until 6 months, and then be through phone support for the remaining 6 months. Warm up and cool down of minimum of five minutes on stationary exercise cycle, rate of perceived exertion (RPE) ~11, followed by gentle stretching. Progressive resistance training (PRT) will use eight PRT machines training large muscle groups (e.g. bench press, latissimus pulldown, bicep curl, triceps pull down, leg press, knee extension, hamstring curl, calf raises). Intensity will be 80% of one repetition maximum (1RM), building up to 3 sets of 8 repetitions. 1RM will be re-assessed monthly, and program adjusted accordingly.
  Arms: Exercise

SUMMARY:
The proposed research aims to examine whether regular aerobic exercise can preserve renal function, improve aerobic capacity, physical and psychosocial function, strength, cardiovascular function, general well-being and quality of life. Ultimately, the research aims to prove that exercise is a more cost-effective and a more efficient use or healthcare resources used in the treatment of patients with CKD. Exercise is a relatively cheap treatment option which is readily available and accessible for this patient population. establish if, compared with usual care, an exercise programme for pre-dialysis CKD patients;

1. Preserves renal function.
2. Improves aerobic capacity, physical and psychosocial function, strength, cardiovascular function, general well-being and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* - Stages 3-4 chronic kidney disease (CKD) patients (glomerular filtration rate (GFR) 20-60 mL/min)
* Male or female
* Aged >18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy

  * Requiring support for ambulation less than 20m
  * Vasculitis,
  * Proliferative diabetic retinopathy,
  * Severe osteodystrophy,
  * Uncontrolled diabetes,
  * Psychiatric illness, including anxiety, mood and untreated eating disorders
  * Infection or course of antibiotics within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
kidney function | up to 12 months
  estimated glomerular filtration rate (egfr) creatinine

SECONDARY OUTCOMES:
Cardio-respiratory fitness testing (VO2peak) | Baseline, 6 and 12 months
  cycle ergometer
Pulse Wave Velocity (arterial stiffness) | Baseline, 6 and 12 months
  Vicorder equipment, carotid-femoral region.
Body mass index (BMI) | Baseline, 6 and 12 months
weight | Baseline, 6 and 12 months
Waist circumference | Baseline, 6 and 12 months
Duke's activity status index | Baseline, 6 and 12 months
  questionnaire
Short Form 36 questionnaire | Baseline, 6 and 12 months
Total cholesterol | Baseline, 6 and 12 months
High sensitivity c-reactive protein (Hs CRP) | Baseline, 6 and 12 months
Blood pressure | Baseline, 6 and 12 months
Resting heart rate (HR) | Baseline, 6 and 12 months
Triglycerides | baseline, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: sharlene greenwood, Bsc, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, London, United Kingdom